CLINICAL TRIAL: NCT00519480
Title: A Two-Week, Randomized, Double-Blind, Repeat-Dose, Parallel-Group Study to Evaluate the Safety and Tolerability of Metformin > 2000mg Co-Administered With Either GSK189075 500mg BID or GSK 189075 750mg BID to Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study To Assess The Safety And Tolerability Of GSK189075 When Given With A Total Daily Dose Of >/ 2000mg of Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KG2110243
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Tolerability; GSK189075,; Metformin,; Safety,; Diabetes,
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subjects receiving treatment P (Placebo Comparator): Eligible subjects will receive placebo twice daily along with metformin twice daily for 13 days.
  Interventions: Drug: Metformin; Drug: Placebo
- Subjects receiving treatment A (Experimental): Eligible subjects will receive GSK189075 500 milligrams twice daily along with metformin twice daily for 13 days.
  Interventions: Drug: GSK189075; Drug: Metformin
- Subjects receiving treatment B (Experimental): Eligible subjects will receive GSK189075 750 milligrams twice daily along with metformin twice daily for 13 days.
  Interventions: Drug: GSK189075; Drug: Metformin

INTERVENTIONS:
Drug: GSK189075 — GSK189075 will be available as an oral tablet with dosing strengths of 500 milligrams and 250 milligrams.
  Arms: Subjects receiving treatment A; Subjects receiving treatment B
Drug: Metformin — Metformin will be available as an immediate release oral tablet with dosing strengths of 500 milligrams and 850 milligrams.
Drug: Placebo — Placebo will be available as an oral tablets.
  Arms: Subjects receiving treatment P

SUMMARY:
This study will assess safety and tolerability of metformin plus GSK189075 in people with Type 2 Diabetes. About 48 people will participate in this study. Volunteers will not know if they are receiving GSK189075 or a placebo. Participation will last about 5 weeks including a run-in period of up to 2 weeks if necessary to increase metformin up to 2000mg daily, a 13-day treatment period, and a follow-up visit about 1 week after the treatment period. Volunteers will remain in the research clinic beginning 2 days before they receive the first dose of GSK189075 until after the morning dose on the fourth day and from the afternoon of the 12th day of dosing until the morning after the last dose. They will have clinic visits on dosing Days 6, 8, and 10. Volunteers will be given equipment and instructions for measuring their blood sugar at home and will be asked to keep a study diary. Blood pressure, heart rate, laboratory tests on blood and urine, physical examinations, reports of drug side effects and ECGs will be obtained during the clinic visits to assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes for at least three months prior to study
* Diabetes treated with metformin only
* Give consent and sign an informed consent form.
* Agree to follow specific requirements of birth control during participation.

Exclusion Criteria:

* Type I Diabetes.
* Treatment with insulin within 3 months prior to screening
* History of diabetic ketoacidosis or lactic acidosis
* Allergy or sensitivity to metformin or similar drugs or any medical conditions which prohibit metformin use
* Excessive blood donation 56 days before the start of the study
* Urinary tract or bladder infections within four weeks of study start
* Alcohol abuse or illicit drug use within 12 months of study start
* Receiving other investigational drugs or participating in other research trials within 30 of the study start
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements with 7-14 days of study start
* Live alone without regular, daily interactions with someone who can be an emergency contact

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09-11 (Actual); Primary Completion 2008-04-01 (Actual); Study Completion 2008-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical laboratory tests, ECGs, physical exam & adverse events: | screening, in-clinic stays, outpatient clinic visits & follow up visit (approximately 50 days)
Home diary of blood sugar results, adverse events and drug dosing. | throughout the study (approximately 50 days)

SECONDARY OUTCOMES:
study drug blood levels: | Dosing Days 1 & 13 metformin blood levels: Days -1 & 13
Blood glucose & insulin levels following oral glucose challenge: | Dosing Days -1 & 13
fluid intake & output | dosing Days -1 - 3, 13

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (2):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, San Antonio, Texas
- GSK Investigational Site, Buenos Aires, Argentina
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Dobbins R, Hussey EK, O'Connor-Semmes R, Andrews S, Tao W, Wilkison WO, Cheatham B, Sagar K, Hanmant B. Assessment of safety and tolerability of remogliflozin etabonate (GSK189075) when administered with total daily dose of 2000 mg of metformin. BMC Pharmacol Toxicol. 2021 Jun 13;22(1):34. doi: 10.1186/s40360-021-00502-0. PMID 34120651
- See also: Results for study KG2110243 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/KG2110243?search=study&study_ids=KG2110243#rs